CLINICAL TRIAL: NCT04171908
Title: Effects of a Semi-inmersive Virtual Reality Training Program on Muscle Strength, Coordination, Fatigue, Functionality and Quality of Life in Patients With Multiple Sclerosis
Brief Title: Semi-inmersive Virtual Reality on Upper Limb in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Full proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Virtual Arms-EM
Record Dates: First submitted 2019-11-12; First posted 2019-11-21 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis; Treatment Adherence; Upper Extremity Paresis
MeSH Terms: conditions — Multiple Sclerosis; Treatment Adherence and Compliance; Paresis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Conventional Physical therapy for the upper limb
  Interventions: Other: Conventional therapy
- semi-inmersive VR technology plus conventional therapy (Experimental): Conventional Physical therapy for the upper limb plus semi-inmersive VR technology
  Interventions: Other: semi-inversive tech

INTERVENTIONS:
Other: Conventional therapy — Conventional Physical therapy for the upper limb
  Arms: Conventional therapy
Other: semi-inversive tech — Conventional Physical therapy for the upper limb plus Semi-inversive tech
  Arms: semi-inmersive VR technology plus conventional therapy

SUMMARY:
Video games based on VR technology are emerging as valid tools used in neurorehabilitation for patients with neurological disorders, and as a low cost and easily accepted adjunct to traditional therapy. Standard games such as the Nintendo Wii, Playstation Move and Kinect plus XBOX 360 have been used in EM rehabilitation. However, often these are either too difficult for patients or the games progress too quickly, failing to provide impairment-focused training or specifically address patients' needs [10]. Therefore, it is necessary to develop specific serious games for EM patients. Serious games are defined as games designed for a primary purpose other than that of pure entertainment, and which promote learning and behavior changes for EM patients. In this context, gesture caption devices (such as MYO, LEAP or Joy Con´s Nintendo Switch), which uses a sensor that captures the movement of the patient's forearms and hands are really interesting in rehabilitation contexts. This generates a virtual image of the upper limbs on a computer screen and the patient is prompted to perform movements according to the functional task proposed. This system presents important advantages namely thanks to its portability, ease of use, commercial availability, low cost and non-invasive nature. However, evidence is lacking that supports the therapeutic use of semi-inmersive VR technology in the treatment of upper limb (UL) motor disorders in EM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to McDonald's criteria.
* Assessment on the Kurtzke Scale of the State of Multiple Sclerosis Disability (EDSS) with a score between 1.0 and 7.5.
* Stable medical treatment for at least six months prior to the intervention.
* Muscle tone in the upper extremities not greater than 2 points (moderate hypertonia, increased muscle tone during most of the arc of movement, but the affected part can easily be moved passively) on the modified Ashworth Scale.
* Score less than or equal to 4 points in the section ¨Piramidal Function¨ of the functional scale of the EDSS.
* Absence of cognitive impairment, with the ability to understand the instructions and obtain a score equal to or greater than 24 in the Minimental Test.
* Score equal to or less than 2 points in the section ¨Functions Mental¨ of the EDSS.

Exclusion Criteria:

* Diagnosis of another neurological disease or musculoskeletal disorder other than MS.
* Diagnosis of any cardiovascular, respiratory or metabolic disease.
* Other conditions that may interfere with this study, having suffered an exacerbation or hospitalization in the last 3 months before starting the protocol of assessment, or during the therapeutic intervention process.
* Having received a steroid cycle, intravenously or orally, 6 months before the start of the assessment protocol and within the intervention period of study duration.
* Having received treatment with botulinum toxin in the six months prior to the start of the study.
* Presence of uncorrected visual disturbances through eye devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Jamar | 8 weeks
  Hand-held dynamometer: it is an instrument to measure the maximumisometric strength of the hand and forearm muscles. It consists of a sealed hydraulic system with adjustable hand spacing that measures hand grip force. The strength reading can be viewed as pounds or kilograms.Thedynamometer is used for testing the hand grip force and for tracking the grip strength improvements during rehabilitation.
Box and blocks | 8 weeks
  Coordination test: to measure unilateral gross manual dexterity in both the less and more affected side. The Box and blocks consists of moving the maximum number of blocks from one compartment of a box to another, one by one, within one minute. The Box and blocks is a quick, simple, and reliable measurement of manual dexterity. Its administration procedure is standardized and its validity has been shown in elderly subjects with upper limb disability
The Purdue Pegboard Test | 8 weeks
  Motricity: to assess coordination, speed of movement and fine motor dexterity. The The Purdue Pegboard Test features a board with two columns with 25 holes each and a specific number of pins, washers and collars placed in four containers across the top of the board. The test consists of inserting as many pins as possible in three distinct phases, with a time limit of 30 s for each. First, the test is performed with the less affected side, then with the more affected side, then with both hands at the same time and, finally, an assembly test is performed (60 s). The number of pins inserted is subsequently recorded.
Nine Hole Peg Test | 8 weeks
  Motricity: It is a hand function test, which consists of a plastic peg board (25.0 cm × 12.7 cm × 2.3 cm) with nine holes (2.54 cm between the holes) and nine pegs (3.2 cm long, 0.64 cm wide). The participant had to put the nine pegs in the peg board as fast as possible, one at the time with one hand only, and remove them again. The test was performed two times per hand, with the non-affected hand first. The time it takes to fulfill the second trial with the more-affected hand was used for the analysis

SECONDARY OUTCOMES:
The Client Satisfaction Questionnaire | after 8 weeks of treatment
  The Client Satisfaction Questionnaire was used to evaluate the satisfaction of health service users for both groups. This is a self-administered post-treatment questionnaire, comprising eight items which evaluate the level of satisfaction regarding the care and quality of the service received and the level of fulfillment of the patient's expectations regarding the treatment administered. The total score of the questionnaire is 32 points, with higher values meaning higher satisfaction with the treatment received
Adherence | after 8 weeks of treatment
  The attendance rate (%) for therapy sessions (compliance) will be registered

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Cano de la Cuerda, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcos-Anton S, Cano-de-la-Cuerda R, Aranda-Reneo I, Jardon-Huete A, Ona-Simbana ED, Oliva-Moreno J. Cost-effectiveness analysis of the MYO Armband(R) device in combination with specifically designed video games for upper limb rehabilitation in people with multiple sclerosis. J Neuroeng Rehabil. 2025 Nov 27. doi: 10.1186/s12984-025-01801-x. Online ahead of print. PMID 41299524
- [Derived] Marcos-Anton S, Jardon-Huete A, Ona-Simbana ED, Blazquez-Fernandez A, Martinez-Rolando L, Cano-de-la-Cuerda R. sEMG-controlled forearm bracelet and serious game-based rehabilitation for training manual dexterity in people with multiple sclerosis: a randomised controlled trial. J Neuroeng Rehabil. 2023 Aug 19;20(1):110. doi: 10.1186/s12984-023-01233-5. PMID 37598176
- [Derived] Cuesta-Gomez A, Martin-Diaz P, Sanchez-Herrera Baeza P, Martinez-Medina A, Ortiz-Comino C, Cano-de-la-Cuerda R. Nintendo Switch Joy-Cons' Infrared Motion Camera Sensor for Training Manual Dexterity in People with Multiple Sclerosis: A Randomized Controlled Trial. J Clin Med. 2022 Jun 7;11(12):3261. doi: 10.3390/jcm11123261. PMID 35743333
- [Derived] Cuesta-Gomez A, Sanchez-Herrera-Baeza P, Ona-Simbana ED, Martinez-Medina A, Ortiz-Comino C, Balaguer-Bernaldo-de-Quiros C, Jardon-Huete A, Cano-de-la-Cuerda R. Effects of virtual reality associated with serious games for upper limb rehabilitation inpatients with multiple sclerosis: randomized controlled trial. J Neuroeng Rehabil. 2020 Jul 13;17(1):90. doi: 10.1186/s12984-020-00718-x. PMID 32660604